CLINICAL TRIAL: NCT01483833
Title: Protocol for the Study of the Effects of S-MPEC (Iferanserin) in Patients With Hemorrhoids
Brief Title: Efficacy Study of Iferanserin to Treat Hemorrhoids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ventrus Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VEN309-SMPEC-001
Record Dates: First submitted 2011-11-22; First posted 2011-12-01 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2011-11

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — iferanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iferanserin (Active Comparator): Iferanserin administration intra-anally twice daily for 14 days
  Interventions: Drug: Iferanserin
- Placebo (Placebo Comparator): Placebo administration intra-anally twice daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iferanserin — Iferanserin 0.5% ointment applied intra-anally twice daily for 14 days
  Other Names: VEN309
  Arms: Iferanserin
Drug: Placebo — Placebo ointment applied intra-anally twice daily for 14 days
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of topical 0.5% S-MPEC cream vs. placebo cream (applied twice daily for 14 days) in the treatment of Grade I - III hemorrhoids.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of grade I - III hemorrhoids with bleeding episodes of at least every other day during the last two weeks before enrollment in the study.
* Patients signing the Informed Consent form.

Exclusion Criteria:

* Patients with protruding or irreducible hemorrhoids (grade IV).
* Patients with anal fistulas, periproctitis or hemorrhagic diathesis
* Patients with current history of Type I or Type II diabetes mellitus.
* Patients with severe hepatic, renal or cardiovascular disorders.
* Patients with any type of infectious disease.
* Patients who have been involved with another experimental drug trial within the past 30 days.
* Patients presently diagnosed with cancer.
* Patients who have known alcohol and drug abuse.
* Patients who require the use of suppositories.
* Patients with blood or urine laboratory values outside the normal limits or those with values considered abnormal in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2001-09; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Assessment of hemorrhoid bleeding | Day 7 and 14
  Change from pre-treatment in patient assessment of hemorrhoid bleeding (10-point scale: 1=Not at all, 10=Extremely) at the end of one- and two-weeks of treatment are the primary efficacy endpoints for the study.

SECONDARY OUTCOMES:
Assessment of bleeding, hemorrhoid size, other hemorrhoid symptoms, and physician evaluation of hemorrhoids. | 14 days
  Change from pre-treatment in patient assessment of bleeding on other treatment days, change from pre-treatment in hemorrhoid size, change from pre-treatment in patient assessment of other hemorrhoid symptoms/conditions on all treatment days, and physician evaluation of hemorrhoids at the end of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Alexander Herold, MD, Mannheim, Germany

REFERENCES:
- [Derived] Herold A, Dietrich J, Aitchison R. Intra-anal Iferanserin 10 mg BID for hemorrhoid disease: a prospective, randomized, double-blind, placebo-controlled trial. Clin Ther. 2012 Feb;34(2):329-40. doi: 10.1016/j.clinthera.2011.12.012. Epub 2012 Jan 11. PMID 22244049